CLINICAL TRIAL: NCT02491723
Title: Macrolide Mediates Pulmonary Infection of Pseudomonas Aeruginosa Via NLRC4 Inflammasome Signaling Pathway
Brief Title: Macrolide Mediates Pulmonary Infection of Pseudomonas Aeruginosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jin-Fu Xu (Other)
Responsible Party: Sponsor-Investigator, Jin-Fu Xu, deputy director, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150619
Record Dates: First submitted 2015-07-03; First posted 2015-07-08 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Azithromycin; Macrolides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azithromycin group (Experimental): Patients with non-cystic bronchiectasis were treated with azithromycin. The intervention was 500mg daily for three to five days.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Patients with bronchiectasis treated with Azithromycin for three to five days.
  Other Names: macrolide

SUMMARY:
It is acknowledged that IL-18, as a product of the inflammasome, is involved in host defence against viral and bacterial stimuli by modulating the immune response. The aim of this study was to determine IL-18 levels in serum of patients with Bronchiectasis and to investigate whether macrolide attenuate its levels.

DETAILED DESCRIPTION:
Non-cystic fibrosis bronchiectasis is a respiratory disease characterized by persistent airway inflammation and dilation of bronchial wall driven by various causes. Patients with bronchiectasis suffer from excessive sputum production, recurrent exacerbations, and progressive airway destruction. It was reported that 30%-40% patients were infected with Pseudomonas aeruginosa. Major therapy for bronchiectasis is focused on breaking the "vicious cycle" of mucus stasis, infection, inflammation, and airway destruction. Currently a number of clinical trials have showed that macrolide effectively used in the treatment of non-CF bronchiectasis. Evidence has indicated that 14- and 15-membered ring macrolides possess immunomodulation and anti-inflammatory functions beyond their antimicrobial properties. However, the underlying mechanisms that account for the anti-inflammatory actions of macrolides have not yet to be elucidated, and the activities do not appear to be controlled by a single mechanism.Interleukin-18 (IL-18), along with interleukin-1b (IL-1b), is produced by inflammasomes when activated by a number of pathogen, environmental or host-derived danger signals. Inflammasomes are innate immune regulatory protein complexes which seem to play a key role in the host immune response of patients with Bronchiectasis. The aim of this study was to determine IL-18 levels in serum of patients with Bronchiectasis and to investigate whether macrolide could attenuate its levels.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent.
2. Confirmed diagnosis of bronchiectasis by HRCT.
3. Aged 18-85 years.

Exclusion Criteria:

1. Bronchiectasis as a result of CF or active tuberculosis or non-tuberculous mycobacterial (NTM) infection.
2. Allergy to macrolide antibiotics
3. Any history of severe cardiopulmonary dysfunction, eg. left heart failure, Unstable cardiac arrhythmias
4. pregnant or nursing
5. hypogammaglobulinemia or other autoimmune disease 6. diagnosed with ABPA

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
IL-18 in plasma | after 3-5 days treatment of Azithromycin immediately

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Fu Xu, PhD, Study Director — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China